CLINICAL TRIAL: NCT04100941
Title: Comparing the Diagnostic Efficacy of Different Suction Techniques for Endoscopic Ultrasound-guided Fine-needle Biopsy of Pancreatic Solid Lesions Using 25G Procore Needle: a Prospective Randomized Controlled Multicentric Clinical Study
Brief Title: Comparing the Diagnostic Efficacy of Different Suction Techniques for EUS-FNB of Pancreatic Solid Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Shenzhen People's Hospital (Other); The Affiliated Hospital Of Southwest Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, chief of the Gastroenterology, Changhai Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: EUS-FNB 25G
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Pancreatic Mass

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard suction (Experimental): This arm will include all the patients that will get an endoscopic ultrasound guided fine needle biopsy done with the standard suction technique with 10ml negative pressure
  Interventions: Diagnostic Test: standard suction
- slow pull (Experimental): This arm will include all the patients that will get an endoscopic ultrasound guided fine needle biopsy done with the slow pull technique
  Interventions: Diagnostic Test: slow pull
- wet suction (Experimental): This arm will include all the patients that will get an endoscopic ultrasound guided fine needle biopsy done with the wet suction technique
  Interventions: Diagnostic Test: wet suction

INTERVENTIONS:
Diagnostic Test: standard suction — After the needle is inserted in the mass, removing the stylet before performing EUS-FNA. Then attach a 10mL syringe to the end of needle. 20 times of for-backward Suction was applied after the lesion was punctured.
  Arms: standard suction
Diagnostic Test: slow pull — After the needle is inserted in the mass, slowly pull the stylet out while performing EUS-FNA with 20 times for-backward.
  Arms: slow pull
Diagnostic Test: wet suction — After removing the stylet, the needle was flushed with 5mL of saline solution to replace the column of air with saline. A 10mL syringe was attached to the end of the needle. 20 times of for-backward Suction was applied after the lesion was punctured.
  Arms: wet suction

SUMMARY:
There are many factors that can affect the diagnostic yield of EUS-FNA, including lesion factors, the endoscoist experience, the needle size, the number of needle passes, and the suction technique. since diagnostic efficacy of different suction techniques for EUS-FNB is still uncertain, thus we decided to compare the diagnostic efficacy of three common methods: the 10 ml standard negative pressure, slow pull and wet suction.

DETAILED DESCRIPTION:
the standard suction: after the needle is inserted in the mass, removing the stylet before performing EUS-FNA. Then attach a 10mL syringe to the end of needle. 20 times of for-backward Suction was applied after the lesion was punctured.

slow-pull : after the needle is inserted in the mass, slowly pull the stylet out while performing EUS-FNA with 20 times for-backward.

wet suction: after removing the stylet, the needle was flushed with 5mL of saline solution to replace the column of air with saline. A 10mL syringe was attached to the end of the needle. 20 times of for-backward Suction was applied after the lesion was punctured.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years,male or female
2. diagnosis or suspection of solid pancreatic mass based on previous imaging examination (ultrasonography, CT or MRI)
3. lesion diameter larger than 1 cm
4. signed informed consent letter

Exclusion Criteria:

1. pregnant female
2. Pancreatic cystic lesions
3. Anticoagulant/antiplatelet therapy cannot be suspended
4. unable or refuse to provide informed consent
5. Coagulopathy (platelet count < 50× 103/μL,international normalized ratio > 1.5)
6. Severe cardiopulmonary dysfunction that cannot tolerate intravenous anesthesia
7. with history of mental disease
8. other medical conditions that are not suitable for EUS-FNB

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of each individual technique | 1 year
  The results are compared with the gold standard and calculated the accuracy
diagnostic sensitivity of each individual technique | 1 year
  The results are compared with the gold standard and calculated the sensitivity
specificity of each individual technique | 1 year
  The results are compared with the gold standard and calculated the specificity

SECONDARY OUTCOMES:
adverse event rate of each individual technique | 1 year
  record any adverse events related to the procedure
adequacy of specimens obtained by each individual technique | 1 year
  the adequacy will be determined by the pathologists analyzing the sample using a pre-defined scale. They will be blinded to the technique used
cellularity | 1 year
  the cellularity will be determined by the pathologists analyzing the sample using a pre-defined scale. They will be blinded to the technique used
blood contamination | 1 year
  the blood contamination will be determined by the pathologists analyzing the sample using a pre-defined scale. They will be blinded to the technique used

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-shen Li, M.D.,Ph.D., Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No